CLINICAL TRIAL: NCT00228969
Title: Safety and Efficacy of 333369 in the Treatment of Partial Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 333369-EPY-2003
Record Dates: First submitted 2005-06-30; First posted 2005-09-29 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Refractory Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — S-2-O-carbamoyl-1-o-chlorophenyl-ethanol

INTERVENTIONS:
Drug: RWJ-333369

SUMMARY:
The primary objective of this study is to evaluate the efficacy, safety, and tolerability of 4 daily doses of RWJ-333369 as adjunctive treatment of refractory partial epilepsy in subjects who are between 18 and 70 years of age, inclusive

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old,
2. Diagnosis of epilepsy for at least 1 year,
3. Presenting, on average, at least 3 partial onset seizures per month,
4. Currently treated with a stable dose (i.e., for at least 4 weeks) of no more than 3 anti-epileptic drugs (AEDs),

Exclusion Criteria:

1. Have experienced status epilepticus in the past 3 months,
2. Have any serious diseases,
3. History of major psychiatric disorders within the past 2 years.
4. Have received an experimental drug/device within the past 30 days
5. Are pregnant or breastfeeding.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (29):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Northport, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Irvine, California
  - Northridge, California
  - Sacramento, California
  - Fort Collins, Colorado
  - Wilmington, Delaware
  - Decatur, Georgia
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Golden Valley, Minnesota
  - Saint Paul, Minnesota
  - Chesterfield, Missouri
  - Cincinnati, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Sellersville, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - El Paso, Texas
  - Bennington, Vermont
  - Charlottesville, Virginia
  - Roanoke, Virginia
  - Madison, Wisconsin
- Argentina (3):
  - Ciudad de Buenos Aires
  - Córdoba
  - Salta
- Hungary (5):
  - Budapest
  - Debrecen
  - Győr
  - Pécs
  - Zalaegerszeg-Pozva
- Netherlands (4):
  - Breda
  - Heemstede
  - Heeze
  - Rotterdam
- Poland (8):
  - Gdansk
  - Katowice
  - Kielce
  - Krakow
  - Lublin
  - Mosina
  - Warsaw
  - Zabrze
- Russia (3):
  - Moscow
  - Saint Petersburg
  - Samara
- Spain (4):
  - Barcelona
  - Madrid
  - Málaga
  - Pamplona
- United Kingdom (5):
  - Glasgow
  - Middlesbrough
  - Northampton
  - Oxford
  - Reading

REFERENCES:
- [Derived] Lu C, Zheng J, Cao Y, Bresnahan R, Martin-McGill KJ. Carisbamate add-on therapy for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2021 Dec 6;12(12):CD012121. doi: 10.1002/14651858.CD012121.pub2. PMID 34870321